CLINICAL TRIAL: NCT06374901
Title: A Multicenter, Prospective Phase II Clinical Study of Tislelizumab in Combination With Chemotherapy for the Perioperative Treatment of Resectable Locally Advanced Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Tislelizumab Combined With Neoadjuvant Chemotherapy Used in the Perioperative Treatment.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiangdong Cheng (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Shanxi Province Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor-Investigator, Xiangdong Cheng, Chief physician, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-311
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (MHC-II positive with Tislelizumab and SOX/XELOX) (Experimental): Preoperative treatment with Tislelizumab and SOX/XELOX for MHC-II positive patient.
  Interventions: Drug: Tislelizumab; Drug: SOX/XELOX
- B (MHC-II positive with SOX/XELOX) (Active Comparator): Preoperative treatment with SOX/XELOX for MHC-II positive patient.
  Interventions: Drug: SOX/XELOX
- C (MHC-II negative with Tislelizumab and SOX/XELOX) (Experimental): Preoperative treatment with Tislelizumab and SOX/XELOX for MHC-II negative patient.
  Interventions: Drug: Tislelizumab; Drug: SOX/XELOX
- D (MHC-II negative with SOX/XELOX) (Active Comparator): Preoperative treatment with SOX/XELOX for MHC-II negative patient.
  Interventions: Drug: SOX/XELOX

INTERVENTIONS:
Drug: Tislelizumab — Preoperative treatment with Tislelizumab
  Arms: A (MHC-II positive with Tislelizumab and SOX/XELOX); C (MHC-II negative with Tislelizumab and SOX/XELOX)
Drug: SOX/XELOX — Preoperative treatment with SOX/XELOX

SUMMARY:
To evaluate the efficacy of Tislelizumab in combination with chemotherapy versus chemotherapy in neoadjuvant treatment of patients with MHC-II positive (IHC≥2+) and locally advanced gastric/gastroesophageal junction adenocarcinoma by evaluating the main pathologic response rate (MPR).

DETAILED DESCRIPTION:
This study is a multicenter, prospective clinical trial aimed at evaluating the efficacy and safety of Tislelizumab combined with chemotherapy in the perioperative treatment of resectable locally advanced gastric and gastroesophageal junction adenocarcinoma.

A study aimed at untreated gastric and gastroesophageal junction adenocarcinoma patients with resectable locally advanced cT3~4aN+M0 or cT4bNanyM0 (according to AJCC 8th edition staging) The study aimed to enroll 134 untreated resectable locally advanced gastric adenocarcinoma and gastroesophageal junction adenocarcinoma patients, with the primary pathological response rate (MPR) as the primary endpoint.

The subjects need to undergo a screening period examination within 21 days before randomization to determine whether they meet the study conditions. Subjects who meet the research criteria will be randomly divided into MHC - Ⅱ positive group (IHC ≥ 2+) and MHC - Ⅱ negative group (IHC 0/1+) based on their MHC - Ⅱ expression. The MHC - Ⅱ positive group (IHC ≥ 2+) will be randomly divided into two groups in a 1:1 ratio, receiving either Tislelizumab combined with chemotherapy (Group A) or chemotherapy (Group B). The MHC - Ⅱ negative group (IHC 0/1+) will be randomly divided into two groups in a 1:1 ratio, receiving either Tislelizumab combined with chemotherapy (Group C) or chemotherapy (Group D). Randomly stratified factors include Lauren classification (intestinal type vs. diffuse type vs. mixed type).

Based on the sample size assumption of this study, the proportion of MHC - Ⅱ positive population in this study should reach at least 50%.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily joined this study and signed an informed consent form;
* Age ≥ 18 years old, ≤ 75 years old
* Pathological diagnosis of gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction
* Patients must be able to provide fresh slices of tumor tissue (FFPE tissue blocks or approximately 15 slides), unstained FFPE slides, and if clinically feasible, fresh biopsy samples will be preferred. If archived samples cannot be obtained, fresh tumor biopsy specimens must be collected during the baseline period, with the same requirements for glass slides as archived tumor tissue
* Clinical staging determined by CT and laparoscopy for curative resection is cT3~4aN+M0 or cT4bNanyM0 for gastric and gastroesophageal junction adenocarcinoma patients (according to AJCC 8th edition staging)
* Have not received anti-tumor treatment (such as surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.)
* Plan to undergo surgical treatment after the completion of neoadjuvant therapy
* Able to swallow pills normally
* ECOG score 0-1 points
* Expected survival time ≥ 12 months
* Normal function of major organs, i.e. meeting the following criteria:The standard for blood routine examination must comply with: (No blood transfusion or blood products within 14 days, no correction using G-CSF or other hematopoietic stimulating factors)，Neutrophil absolute count ≥ 1.5 × 109/L; Platelets ≥ 80 × 109/L; Hemoglobin ≥ 80g/L
* Biochemical examination must meet the following standards: Total bilirubin<1.5

  * ULN; ALT and AST ≤ 2.5 × ULN; Serum Cr ≤ 1.5 x ULN or endogenous creatinine clearance rate>50ml/min (male: endogenous creatinine clearance rate=(140 age) x body weight)/(72 x serum Cr); Female: Endogenous creatinine clearance rate=(140 age) x body weight/(72 x serum Cr) x 0.85; Weight unit: kg; Serum Cr unit: mg/mL
* Female subjects with pregnancy ability must undergo a serum pregnancy test within 7 days before the first medication, and the result is negative. They are willing to use efficient contraception methods during the trial period and 120 days after the last dose. For male subjects whose partners are women of childbearing age, surgical sterilization or agreement to use efficient methods of contraception during the trial period and 120 days after the last dose should be considered

Exclusion Criteria:

* There are non resectable factors, including tumor reasons that cannot be resected or surgical contraindications that cannot be resected or those who refuse surgery
* Previously or currently suffering from other malignant tumors
* Suffering from any chronic or major illness that is considered intolerable to treatment (such as severe heart disease, uncontrolled hypertension, certain degrees of liver and kidney dysfunction, etc.)
* Those who have experienced gastrointestinal perforation, abdominal abscess in the past, or recent (within 3 months) intestinal obstruction or imaging and clinical symptoms indicating accompanying intestinal obstruction
* If there are significant clinically significant bleeding symptoms or clear bleeding tendencies, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis, within the first 3 months prior to the first use of the study drug, and if fecal occult blood is positive during the baseline period, a follow-up examination can be conducted. If the results are still positive after the follow- up examination, a gastroscopy examination is required (excluding those who have undergone gastroscopy examination within 3 months prior to enrollment to exclude such situations)
* If the patient is in the active infection stage and needs treatment (such as using antibiotics, antiviral drugs, or antifungal drugs)
* Active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU/ml; hepatitis C reference: HCV antibody positive and HCV copy number>upper limit of normal value)
* Patients with congenital or acquired immune dysfunction (such as HIV infected individuals)
* Patients with any active autoimmune diseases or a history of autoimmune diseases with the possibility of recurrence
* Planned or previously received organ or allogeneic bone marrow transplantation
* Subjects who currently have interstitial pneumonia or interstitial lung disease, or have a history of requiring hormone therapy for interstitial pneumonia or interstitial lung disease, or those whose screening period CT shows active pneumonia or severe lung function impairment; Active pulmonary tuberculosis
* Current or recent use of immunosuppressive drugs or systemic corticosteroids for the purpose of achieving immunosuppression
* Patients who have received attenuated live vaccines within 28 days prior to the first use of the study drug, or who need to receive such vaccines during treatment or within 60 days after the last dose
* Known to be allergic to any investigational drug or excipient
* Lactating women
* Any factors determined by the researcher that may affect patient safety and result in the forced termination of this study midway

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
MRP (Main pathological response) | After operation about 2 weeks until postoperative pathology report come out.
  The percentage of subjects who showed no residual tumor cells (including lymph nodes, stage ypT0N0M0) and only residual single or small focal cancer cells under the light microscope

SECONDARY OUTCOMES:
pCR (pathologic complete response) | After operation about 2 weeks until postoperative pathology report come out.
  The percentage of subjects with a TRG grade of 0 who do not have live tumor cell residues in the primary tumor lesion
DFS (Disease free survival) | From date of randomization until the date of first documented progression， assessed up to 100 months
  Refers to the time between the time of baseline imaging evaluation and disease recurrence or death (whichever occurs first) in disease-free subjects after surgery.
OS (Overall survival) | From date of randomization until the date of death, assessed up to 120 months
  The time between the date of enrollment and death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No